CLINICAL TRIAL: NCT03356496
Title: Preoperative Self-managed Respiratory Therapy for Reduction of Postoperative Pulmonary Complications After Non-cardiothoracic Surgery
Brief Title: Preoperative Self-managed Respiratory Therapy for Reduction of Postoperative Pulmonary Complications
Acronym: PRESMART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays due to COVID, standard of care has changed, eliminating the need for the study
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Hari Paudel, Assistant Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO00030057
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Respiratory Complication

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Patient provided with instructions and video for the use of an incentive spirometry device. Patient instructed to use incentive spirometry device as frequently as every hour while awake but at least 4 times daily for at least 10 breathing cycles for 1-3 weeks before surgery. Patient instructed to record usage and any physical complaints in a diary.
  Interventions: Device: AirLife 4000 cc incentive spirometry device
- Control (No Intervention): Patient receives only usual care as provided by perioperative healthcare providers.

INTERVENTIONS:
Device: AirLife 4000 cc incentive spirometry device — Incentive spirometry device provides improved lung expansion and respiratory muscle strength
  Arms: Intervention

SUMMARY:
Postoperative pulmonary complications (PPCs) are a source of much morbidity and mortality. Rates of PPCs exceed 30% in patients with multiple risk factors. Several studies have demonstrated reduced PPCs in patients who underwent preoperative inspiratory muscle training. These studies largely focused on cardiothoracic surgery and required the use of respiratory therapists. The investigators hypothesize that preoperative, self-administered respiratory therapy would reduce PPCs in patients with risk factors for PPCs undergoing any non-cardiothoracic surgery. This study is a randomized, controlled trial comparing preoperative use of an incentive spirometry device with usual care in patients undergoing non-emergent, non-cardiothoracic surgical procedures under general anesthesia.

DETAILED DESCRIPTION:
Postoperative pulmonary complications account for >50% of all adverse postoperative events and are more costly and carry greater comorbidity than cardiac complications. Much research has been performed to identify potential risk reduction strategies for PPCs. Until recently all of these focused on intraoperative and postoperative interventions, including lung-protective mechanical ventilation, lung expansion techniques, and use of regional anesthesia and analgesia. In the last few years several studies have investigated the potential role of preoperative interventions to improve respiratory status. These studies have demonstrated benefit from preoperative inspiratory muscle training (IMT). A recent systematic review found that any preoperative intervention, such as education, IMT, exercise training or relaxation reduced PPC rates. However, these studies have focused on cardiothoracic and abdominal surgery, and almost all have utilized respiratory therapist-directed interventions. Likely due to the additional costs and difficulty of arranging respiratory therapy on an outpatient basis, this promising new risk mitigation strategy has yet to be adopted on a large scale. Incentive spirometry devices offer a potentially easier and less costly preoperative respiratory intervention. Incentive spirometers are a drug-free, easy to use, hand-held device that promotes deep breathing and respiratory muscle strength by providing visual feedback during sustained inhalation. It opens weak or collapsed airways to mobilize and assist mucociliary clearance to the upper airways where it can be coughed out. This study evaluates the hypothesis that providing preoperative, patient self-directed respiratory therapy with use of an incentive spirometry device will reduce the incidence of PPCs in patients with increased pulmonary risk undergoing any major, non-cardiothoracic surgery with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate or high risk for postoperative pulmonary complications as defined by ARISCAT score >25
* Undergoing non-cardiothoracic surgery scheduled at least 7 days in the future
* Planned general anesthesia (alone or in combination with regional or neuraxial anesthesia)
* Personal internet access

Exclusion Criteria:

* Active bronchospasm during preoperative clinic visit
* History of pneumothorax
* History of tracheal stoma or ventilator dependency
* Pregnancy
* Chronic oxygen requirement
* Deficient motor and/or visual function that will prohibit utilization of the device or instructional video and handout
* Lack of English language proficiency
* Inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Up to 30 days after surgery
  Composite of hypoxemia (pulse oximetry <88% with provision of oxygen therapy beyond 24 hours after surgery); bronchospasm (new wheezing or bronchospasm with provision of bronchodilator therapy); hypercarbia (serum bicarbonate or arterial or end-tidal carbon dioxide level above reference range treated with provision of mechanical ventilation); atelectasis (radiographic evidence of atelectasis plus respiratory symptoms or abnormal lung exam findings); respiratory infection (patient received antibiotics for suspected respiratory infection and had at least 1 of following: new or changed sputum, new or changed lung opacities on chest radiograph, fever, or leukocyte count >12,000/microliter); pleural effusion (radiographic evidence of pleural effusion and performance of thoracentesis); pneumothorax (radiographic evidence of pneumothorax); and ventilatory failure (replacement of endotracheal tube or mechanical ventilation for >48 hours postoperatively)

SECONDARY OUTCOMES:
Mortality | Up to 30 days after surgery
  Patient death from any cause
Length-of-stay | Up to 30 days after surgery
  Number of days of hospitalization after index surgery
Readmission | Up to 30 days after surgery
  Incidence of rehospitalization after index surgery
Unanticipated hospital admissions | Up to 30 days after surgery
  Incidence of inpatient admission after index surgery that was planned as outpatient
Unanticipated hospital observation | Up to 30 days after surgery
  Incidence of admission for observation for recovery after index surgery planned as outpatient
Unanticipated intensive care unit utilization | Up to 30 days after surgery
  Incidence of intensive care admission after index surgery not planned for intensive care unit admission

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canet J, Gallart L, Gomar C, Paluzie G, Valles J, Castillo J, Sabate S, Mazo V, Briones Z, Sanchis J; ARISCAT Group. Prediction of postoperative pulmonary complications in a population-based surgical cohort. Anesthesiology. 2010 Dec;113(6):1338-50. doi: 10.1097/ALN.0b013e3181fc6e0a. PMID 21045639
- [Background] Katsura M, Kuriyama A, Takeshima T, Fukuhara S, Furukawa TA. Preoperative inspiratory muscle training for postoperative pulmonary complications in adults undergoing cardiac and major abdominal surgery. Cochrane Database Syst Rev. 2015 Oct 5;2015(10):CD010356. doi: 10.1002/14651858.CD010356.pub2. PMID 26436600